CLINICAL TRIAL: NCT05002933
Title: A 6-month, Multicenter, Prospective, Single-arm, Open-label, Phase IV Study Evaluating the Clinical Efficacy and Safety of Insulin Glargine U300 in Chinese Adult Patients With Uncontrolled Type 2 Diabetes Mellitus With a 3-month Extension Period
Brief Title: A Clinical Efficacy and Safety Study of Insulin Glargine U300 in Chinese Adult Patients With Uncontrolled Type 2 Diabetes Mellitus With a 3-month Extension Period
Acronym: INITIATION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16585; U1111-1251-4484 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insulin glargine 300 U/ml (Experimental): Insulin glargine 300 U/ml once daily for 24 weeks. Participants may continue for an additional 12 week extension period or switch to other anti-diabetic treatment, insulin dose will be adjusted according to the recommended dose titration algorithm
  Interventions: Drug: Insulin glargine 300 U/ml

INTERVENTIONS:
Drug: Insulin glargine 300 U/ml — Solution for injection Subcutaneous injection
  Other Names: HOE901 Toujeo

SUMMARY:
This is a prospective, interventional, single arm, multicenter, phase 4 study to evaluate the clinical efficacy and safety of initiating Insulin glargine U300 in insulin-naive patients or switching from any other basal insulin to Insulin glargine U300 in insulin pre-treated patients with uncontrolled T2DM.

DETAILED DESCRIPTION:
Maximum study duration per participant will be approximately 37 weeks per patient: up to 1 week screening period, 24 weeks insulin glargine U300 treatment period and 12 weeks observational extension period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age≥18 years) who diagnosed with type 2 diabetes
* Patients who should initiate Insulin glargine U300 treatment following local label and guideline at investigator's discretion, including:

  * insulin naive patients (no current or previous insulin used during the last year prior to screening except for a maximum 10 days in relation to acute illness or surgery, etc.) uncontrolled (HbA1c between 7.5% and 11.0%) at screening visit on stable dose treatment with ≤ 2 OADs (metformin, sulfonylurea, thiazolidinedione, DPP-4 inhibitor, SGLT-2 inhibitor, glinide, α-glucosidase inhibitor) within 8 weeks prior to screening, at least one of which must be on maximum tolerated dose, or
  * patients uncontrolled (HbA1c between 7.5% and 11.0%) at screening visit with other basal insulin, or
  * patients controlled with other basal insulin but experienced frequent hypoglycemia or with increased hypoglycemia risk at investigator's discretion
* Patients who treated with basal insulin must have a stable dose of antidiabetic drugs (dose change no more than ±20% vs. the dose on screening visit for basal insulin) within 8 weeks prior to screening

Exclusion Criteria:

* Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening, or at baseline, or any major systemic disease resulting in short life expectancy that in the opinion of the Investigator would restrict or limit the patient's successful participation for the duration of the study
* Use of any product containing short or rapid acting insulin in the last 3 months prior to screening (unless used for ≤10 days in relation to hospitalization or an acute illness)
* Use of oral anti-diabetic drugs other than those allowed and listed in the inclusion criteria, Glucagon-like peptide-1 (GLP-1) receptor agonists, or any investigational agent (drug, biologic, device) within 3 months prior to screening visit
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for two weeks or more within 8 weeks prior to the time of screening
* Known hypersensitivity / intolerance to insulin glargine or any of its excipients
* Pregnant or lactating women
* Women of childbearing potential with no effective contraceptive method
* Participation in another clinical trial

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c from baseline to week 24 | Baseline to Week 24

SECONDARY OUTCOMES:
Mean change in HbA1c from baseline to week 12 and week 36 | Baseline to Week 12 and 36
Percentage of participants achieving HbA1c target <7% | at Week 12, 24 and 36
Percentage of participants achieving HbA1c target <7% without hypoglycemic events | at Week 12 and 24
Mean change in Fasting Plasma Glucose (FPG) from baseline to week 12, 24 and 36 | Baseline to Week 12, 24 and 36
Mean change in fasting Self-Monitored Blood Glucose (SMBG) from baseline to week 12 and week 24 | Baseline to Week 12 and 24
Mean change in of 7-points SMBG per time point from baseline to week 12 and week 24 | Baseline to Week 12 and 24
Mean change in Insulin glargine U300 dose from baseline to week 12, 24 and 36 | Baseline to Week 12, 24 and 36
Number of participants experiencing hypoglycemia from baseline to week 12, 24 and 36 | Baseline to Week 12, 24 and 36
Number of hypoglycemic events per patient-year | Baseline to Week 12, 24 and 36
Number of participants with adverse events | Baseline to Week 24 and 36
Mean change in body weight from baseline to Week 12 and Week 24 | Baseline to Week 12 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Sites, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16585 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25284&tenant=MT_SNY_9011